CLINICAL TRIAL: NCT04872361
Title: Ultrasonographic Assessment of Atelectasis in Major Upper Abdominal Surgeries With Different Ventilatory Strategies
Brief Title: Which Ventilatory Strategy is Better for Lung in Upper Abdominal Surgeries?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MFM-IRB.MD.21.01.412
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia Induced Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind (Participant, Outcomes Assessor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low PEEP (Placebo Comparator): Low positive end-expiratory pressure (PEEP) and no recruitment maneuver (RM)
  Interventions: Procedure: Low PEEP; Device: Lung ultrasonogrphy assessment
- High PEEP (Active Comparator): High positive end-expiratory pressure (PEEP)
  Interventions: Procedure: High PEEP; Device: Lung ultrasonogrphy assessment
- High PEEP/RM (Active Comparator): High positive end-expiratory pressure (PEEP) and recruitment maneuver (RM)
  Interventions: Procedure: High PEEP/RM; Device: Lung ultrasonogrphy assessment

INTERVENTIONS:
Procedure: Low PEEP — Patients will be ventilated with a PEEP of 4 cm H2O and no RMs throughout the study
  Arms: Low PEEP
Procedure: High PEEP — PEEP of 10 cm H2O will be applied
  Arms: High PEEP
Procedure: High PEEP/RM — PEEP of 10 cm H2O and RM (30 cm H2O for 30 s) immediately after the second lung ultrasonographic examination and repeated every 30 minutes till emergence
  Arms: High PEEP/RM
Device: Lung ultrasonogrphy assessment — The thorax will divided into 12 quadrants, each of them will be assigned a score of 0-3 as 0, normal lung sliding with fewer than three single B lines
  1. three or more B lines
  2. coalescent B lines
  3. consolidated lung. The LUS (0-36) will be calculated with higher scores indicating more aeration loss

SUMMARY:
Ventilated Patients especially those undergoing upper abdominal surgeries are prone to lung atelectasis. They are at risk of adverse effects secondary to inadequate lung ventilation.

Applied PEEP and Recruitment maneuver are thought to enhance lung aeration under general anesthesia which could be assessed by ultrasound.

DETAILED DESCRIPTION:
The aim of our study is to assess the effect of using PEEP with and without recruitment maneuver on atelectasis and lung aeration during open upper abdominal surgeries by ultrasonography.

Application of PEEP improves intraoperative oxygenation and thus could minimize the incidence of postoperative atelectasis and respiratory complications during abdominal surgeries.

A recent study found that PEEP and RM prevented intraoperative aeration loss, which didn't persist after extubation when comparing effects of positive end-expiratory pressure/recruitment maneuvers with zero end-expiratory pressure on atelectasis during open gynecological surgery by ultrasonography

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' physical status grades I, II, and III.

Exclusion Criteria:

* Patient refusal.
* Psychiatric diseases.
* Body Mass Index > 35 Kg/m2.
* Previous intrathoracic procedures.
* History of severe obstructive pulmonary disease.
* History of severe restrictive lung disease.
* Pulmonary arterial hypertension ( systolic pulmonary arterial pressure >40 mmHg).
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Pre-emergence LUS score | intraoperative before recovery from anesthesia
  Lung ultrasonography score (LUS score) between groups at the end of surgery (just before emergence) as a lower LUS indicates better lung aeration.

SECONDARY OUTCOMES:
Lung ultrasonography score (LUS score) | preoperative, intraoperative for anesthesia duration to 1 hour postoperative
  Lung ultrasonography score (LUS score) between groups
Heart rate | preoperative, intraoperative for anesthesia duration to 1 hour postoperative
  heart rate between groups at each time point of LUS score performance
Mean blood pressure | preoperative, intraoperative to 1 hour postoperative
  mean arterial blood pressure between groups at each time point of LUS score performance
oxygen saturation | preoperative, intraoperative to 1 hour postoperative
  patient oxygen saturation between groups at each time point of LUS score performance
End-tidal carbon dioxide tension | intraoperative for anesthesia duration
  end tidal CO2 between groups post induction, post recruitment and before extubation
Arterial partial pressure of oxygen (PaO2) | Intraoperative and 15 min postoperative
  arterial blood gases post induction, before extubation and at the PACU
Arterial partial pressure of carbon dioxide (PaCO2) | Intraoperative and 15 min postoperative
  arterial blood gases post induction, before extubation and at the PACU
PaO2/FiO2 | Intraoperative and 15 min postoperative
  arterial blood gases post induction, before extubation and at the PACU
Peak inspiratory pressure | intraoperative for anesthesia duration
  peak inspiratory pressure between groups after intubation
Postoperative pulmonary complications (PPCs) | 5 days
  PPCs include (pneumothorax, pleural effusion, pulmonary collapse, atelectasis, pneumonia, acute respiratory distress syndrome (ARDS), or pulmonary aspiration).

CONTACTS AND LOCATIONS:
Overall Officials: Aboelnour E Badran, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Hanaa M EL- Bendary, MD, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be available after completing the study and acceptance for publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completing the study and acceptance for publication
Access Criteria: Sharing Criteria: the data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients.